CLINICAL TRIAL: NCT06722833
Title: Investigation of Pain, Function and Audiovestibular System Features in Individuals With Temporomandibular Joint Dysfunction
Brief Title: Physiotherapy Investigation in Patient With Temporomandibular Joint Dysfunction
Status: Not yet recruiting | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, FİLİZ EYÜBOĞLU, PhD, Uskudar University
Other Study IDs: tmjstudy1
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: temporomandibular dysfunction; pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Knowing the associated factors for people suffering from TMD may help to develop preventive, therapeutic and health strategies. The aim of this study was to present the assessments of audiovestibular symptoms in people with TMD. The main question it aims to answer is the questions are as follows:

1. Is there a relationship between TMJ symptoms and audiovestibular assessment in people with TMD?

Participants will:

Participants diagnosed with TMD will be informed about the study and informed consent will be obtained. Data obtained after the TMJ and vestibular system evaluation of the participants will be analyzed.

DETAILED DESCRIPTION:
Temporomandibular dysfunction (TMD) is a health condition affecting the temporomandibular joint (TMJ) and related structures. The prevalence of TMD in adults affects a very large portion of the world's population. TMD is complex and multifactorial due to its etiology with neuromuscular, traumatic, degenerative and sociodemographic aspects. The aim of this study is to reveal audiovestibular assessments in individuals with TMD. After obtaining voluntary consent forms, participants are subjected to assessments. The "Statistical Package for Social Sciences (SPSS) Statistics 23.0 (SPSS Inc, Chicago, USA) program will be used in the analysis of the study data. Before starting the analysis of the data, the Kolmogorv Smirnov test will be used to check whether the data is suitable for normal distribution. Data that are suitable for normal distribution will be analyzed with parametric tests, and those that are not suitable for normal distribution will be analyzed with non-parametric tests. Descriptive statistics for quantitative variables will be shown as mean and standard deviation, and for qualitative variables determined by counting, descriptive statistics will be shown as numbers and percentages. T-test/chi square/Mann Whitney U will be used in two-group comparisons, and one-way variance analysis/Kruskal Wallis test will be used in three-group comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study between the ages of 18-35
* Diagnosed with unilateral TMJ disorder at least 1 month ago according to the - Research Diagnostic Criteria of Temporomandibular Disorders (RDC/TMD) classification (Dworkin et al., 1992)
* Having muscle tenderness and pain in the temporomandibular joint region

Exclusion Criteria:

* Traumatic injuries in the same area other than TMD
* Ear diseases that cause hearing loss
* Dentofacial Anomalies
* Receiving orthodontic treatment
* Neurological diseases, vestibular or visual problems

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Young adults diagnosed with TMD
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 1 day (The evaluation will be done one-time)
  Visual analog scale (VAS) will be used to assess the pain intensity of individuals related to TMJD. The individual will be asked to mark the perceived pain intensity on a 10 cm long horizontal line. The individual's pain intensity will be recorded by measuring the distance the individual marks on the line in millimeters.
Evaluation of Temporomandibular Joint Functional Status | 1 day (The evaluation will be done one-time)
  Mandibular Dysfunction Questionnaire (MFBA) was administered to individuals to assess the functional status of the joint and the level of functional impairment that its dysfunction may cause.

SECONDARY OUTCOMES:
Measurement of Temporomandibular Joint Mobility | 1 day (The evaluation will be done one-time)
  Individuals will be instructed to open their mouths as wide as possible without causing pain and joint mobility will be measured and recorded using a millimetric ruler. TMJ movements in all directions will be measured three times and the average of the measurements will be recorded and noted.
Immittancemetric Evaluation | 1 day (The evaluation will be done one-time)
  Before tympanometric evaluation, otoscopic examination is performed. Tympanometry, acoustic reflex and eustachian tube function tests are performed with the Interacoustics® Titan Handheld (Denmark) device.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Eyüboğlu, PhD, Principal Investigator — Uskudar University